CLINICAL TRIAL: NCT05967000
Title: Evaluating a Preventive Heart Health Programme for Perimenopausal Women - Empowering Sustainable Healthy Habits Through Behaviour Change Strategy.
Brief Title: Evaluating a Preventive Heart Health Programme for Women at Midlife
Acronym: Phenomenon
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Alexandra Hospital (Other)
Collaborators: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Other Study IDs: 2022/00350; NUS/BISI/SG02/2022 (Other Grant/Funding Number: NUS)
Record Dates: First submitted 2023-06-30; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Cardiovascular Disease; Menopause
Keywords: preventive cardiology; menopause; implementation
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women at midlife: Women aged 45-65 years with risk factors or pre-existing CVD
  Interventions: Other: Preventive heart health and menopause programme

INTERVENTIONS:
Other: Preventive heart health and menopause programme — This is a one-stop women's heart and menopausal service in a public hospital led by cardiologists and gynaecologists with a multidisciplinary team. Pre-existing speciality care and services are repackaged, and clinic workflows are reworked to provide more streamlined, convenient, and integrated care. Services encompass:
  * Individualised risk assessment, screening, diagnosis, and treatment of CVD.
  * Lifestyle education, adjustment, stress management, and counselling.
  * Smoking cessation programs.
  * Bone health screening, mammogram with access to our co-located gynaecologists and hormone replacement therapy.
  * Virtual consults and health coaching.

SUMMARY:
This study examines the factors that limit or support the implementation of a pilot heart health program for perimenopausal women. The investigators evaluate the effectiveness of this program in raising awareness and promoting behavior change to maintain cardiovascular health.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the leading cause of mortality among women. Heart-related conditions are responsible for the death of one out of every three women. In Singapore, CVD in women causes more morbidity and mortality than breast and cervical cancer. The burden will be exacerbated by Singapore's aging population and the longer life expectancy of women compared to men. Primary and secondary prevention strategies are implemented to reduce the overall impact of CVD on public health. Women who have traditional risk factors are at a greater risk of experiencing heart attacks compared to men with comparable risk factors. Additional risks specific to women include a history of pregnancy complications, breast cancer, and premature menopause. CVDs in women are frequently overlooked in terms of diagnosis and treatment.

Menopause is a phase in a woman's life that brings about significant changes to both her reproductive organs and her physical and psychological well-being. Management issues encompass a spectrum of concerns, including immediate symptoms like insomnia and palpitations, intermediate concerns related to bone health, and long-term considerations associated with the development of cardiovascular disease. The American Heart Association (AHA) provides guidelines for multidisciplinary care aimed at preventing cardiovascular disease (CVD) in women. Countries like Canada have established specialized organizations to address this issue. Collaborative clinics involving cardiologists, gynecologists, and women's heart centers are crucial, even for women who are generally healthy.

The objective of this study is to examine the factors that limit or support the implementation of a preventive heart health program for perimenopausal women. Additionally, the investigators aim to evaluate the effectiveness of our pilot women's health program in raising awareness and promoting behavior change to maintain cardiovascular health.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 45-65 years at risk for cardiovascular disease or with pre-existing cardiovascular disease.
* English speaking

Exclusion Criteria:

* Pregnant women
* Unable to provide informed consent
* Women out of the menopause transition phase of 45-65 years of age.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women going through the menopause transition with risk factors for CVD or pre-existing CVD.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Reach of the programme | 1 year
  This a part of the RE-AIM comprehensive method for programme evaluation. This is measured via participation rate which is the number of eligible women recruited (numerator) divided by the number of eligible women screened for the programme (denominator
Effectiveness of the programme | 1 year
  This a part of the RE-AIM comprehensive method for programme evaluation. This is measured via the GPAQ (Global physical activity questionnaire)
Effectiveness of the programme | 1 year
  This a part of the RE-AIM comprehensive method for programme evaluation. This is measured via the Utian Quality of life scale.
Adoption of the programme | 1 year
  This a part of the RE-AIM comprehensive method for programme evaluation. This is measured via qualitative interviews to assess whether healthcare providers are accepting of the intervention and can sustain the change.
Implementation of the programme | 1 year
  This will be measured as counts from clinic visits

SECONDARY OUTCOMES:
Anthropometric measurements | 1 year
  Weight and height will be combined to report BMI in kg/m^2
Blood pressure | 1 year
  Office blood pressure measurements
Blood biomarkers | 1 year
  Hba1c
Blood biomarkers | 1 year
  Lipid profile
Blood biomarkers | 1 year
  Vitamin D levels
Surveys | At the end of the study at 1 year
  Semi structure interviews will be conducted and analysed via reflexive thematic approach.

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandra Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No